CLINICAL TRIAL: NCT01252758
Title: A Phase II Study to Assess the Efficacy and Safety of a Single Inhaled Dose of Albuterol Sulfate Dry Powder Via the Trivair Deposition System Versus Albuterol Sulfate HFA pMDI in Patients With Intermittent or Persistent Mild Asthma
Brief Title: Dose Finding Study of Albuterol Sulfate in Patients With Intermittent or Persistent Mild Asthma
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Acerus Pharmaceuticals Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: TBS-7-2010-01
Record Dates: First submitted 2010-12-01; First posted 2010-12-03 (Estimated); Last update posted 2018-03-13 (Actual); Status verified 2018-03

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Albuterol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- albuterol sufate DPI (TBS-7) dose 1 (Experimental)
  Interventions: Drug: albuterol sufate DPI (TBS-7) dose 1
- albuterol sufate DPI (TBS-7) dose 2 (Experimental)
  Interventions: Drug: albuterol sufate DPI (TBS-7) dose 2
- albuterol sufate DPI (TBS-7) dose 3 (Experimental)
  Interventions: Drug: albuterol sufate DPI (TBS-7) dose 3
- placebo (Placebo Comparator)
  Interventions: Other: Placebo
- Ventolin HFA dose 1 (Active Comparator)
  Interventions: Drug: Albuterol
- Ventolin HFA dose 2 (Active Comparator)
  Interventions: Drug: Albuterol

INTERVENTIONS:
Drug: albuterol sufate DPI (TBS-7) dose 1
  Arms: albuterol sufate DPI (TBS-7) dose 1
Drug: albuterol sufate DPI (TBS-7) dose 2
  Arms: albuterol sufate DPI (TBS-7) dose 2
Drug: albuterol sufate DPI (TBS-7) dose 3
  Arms: albuterol sufate DPI (TBS-7) dose 3
Other: Placebo
  Arms: placebo
Drug: Albuterol
  Arms: Ventolin HFA dose 1
Drug: Albuterol
  Arms: Ventolin HFA dose 2

SUMMARY:
The drug product albuterol sulfate DPI, TBS-7, is a single dose inhalation product of albuterol sulfate containing 240 ug albuterol sulphate (200 ug of albuterol) and inhalation grade lactose in a new dry powder delivery system called the Trivair deposition system.

Three different doses of albuterol sulfate DPI, TBS-7, will be administered in this dose ranging clinical trial: an optimal dose, 80% of the optimal dose and 50% of the optimal dose and will be compared with placebo and an active comparator.

ELIGIBILITY:
Inclusion Criteria:

1. Generally healthy male or female subjects, over the age of 18. Females of child bearing potential must be non-pregnant (confirmed by a negative serum hCG test at the screening visit) or non-lactating.
2. Documented clinical history (minimum six months) of intermittent or mild persistent asthma according to the Global Initiative for Asthma (GINA, 2009) criteria requiring and responding to short acting inhaled b2-agonist (SABA) therapy.
3. Using a SABA alone, or concurrent use of anti-inflammatory therapy, (i.e. Singulair,® theophylline or inhaled corticosteroid (ICS)). The dose and frequency of anti-inflammatory medication should be stable for at least four weeks prior to the screening visit. For subjects who are currently taking an ICS, the total daily dose should not exceed 1000µg budesonide or equivalent steroid.
4. A pre-bronchodilator FEV1 ≥ 60% to 90% of predicted at screening.
5. Confirmed diagnosis of asthma by demonstrating: Reversibility of airway obstruction of ≥ 12% increase in FEV1 within 30 minutes after the inhalation of a standard dose of albuterol (2 puffs, 180 µg) delivered via pMDI.
6. Nonsmokers or ex-smokers (stopped at least 6-month period prior to the screening visit).

Exclusion Criteria:

1. A change in asthma mediation within the previous four weeks of screening visit.
2. A life-threatening asthma episode within the last six months or > 2 within the past year. A life-threatening asthma episode is defined as an asthma exacerbation which required hospitalization and/or was associated with hypercapnia, respiratory arrest, or hypoxic seizures.
3. If in the Investigator's opinion, the subjects asthma severity is too severe to participate in the study, or they would be unable to withhold their asthma medication for the times outlined above as well as require the use of daily high dose ICS (>1000µg budesonide or equivalent).
4. Use of a long acting inhaled b2-agonist (LABA), ipratropium bromide containing medication (ie. Combivent) or Tiotropium therapy.
5. Use of any oral, depot or parental corticosteroids within four weeks of screening visit. The use of topical corticosteroid cream (<1%) to treat skin conditions is allowed.
6. History of an upper or lower respiratory tract infection requiring antibiotics; emergency room treatment in the preceding four weeks; or hospitalization in the previous three months; or a history of multiple hospital visits for treatment of their respiratory disease.
7. History of any immediate or delayed hypersensitivity reaction to inhaled b2-agonists, lactose, milk-protein, or excipients (pMDI inhalers) any component of the formulations.
8. Clinically significant history or current evidence of any of the diseases listed below. Clinically significant is defined as any diseases that in the opinion of the Investigator would put the subject at risk through study participation. These include, but are not limited to:

   * bronchiectasis, bronchopulmonary dysplasia, cystic fibrosis, emphysema, chronic bronchitis, or other significant lung diseases
   * hypertension which, in the opinion of the Investigator, deems the subject unfit to enter the study; subjects must not have a persistent systolic pressure above 145 mmHg or diastolic pressure above 85 mmHg unless the Investigator confirms that it is satisfactory for their age.
   * arrhythmias, coronary artery disease, congestive heart failure, congenital heart disease or other significant cardiac disease
   * diabetes mellitus requiring medication
   * cirrhosis, alcoholism, biliary obstruction or other hepatic disease
   * epilepsy, psychosis, or other conditions/diseases of the nervous system
   * malignancy
   * current or past history of glaucoma
9. Clinically significant ECG abnormalities.
10. History of seasonal allergic rhinitis that would require treatment during the study period.
11. History of immunotherapy within six months of the screening visit or planned initiation of immunotherapy within the study period. Subjects will be allowed to enter the study if undergoing de-sensitization to a specific allergen for at least six months on a stable maintenance dose prior to the screening visit. Seasonal pollen de-sensitization therapy is allowed if this is not the initial course and no significant adverse effect was observed with the previous administration.
12. Laboratory value exceeding the limit of normal and determined to be clinically relevant by the Investigator.
13. Use of concomitant medications which might interfere with participation in the study or the interpretation of data.
14. Current smokers.
15. Known or suspected history of alcohol drug or drug/solvent abuse

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-11; Primary Completion 2013-04 (Estimated); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
forced expiratory volume at one second | 6 hours

SECONDARY OUTCOMES:
PK parameters | 6 hours
safety and tolerability | 7 days